CLINICAL TRIAL: NCT00508209
Title: Phase II Study of Bortezomib Dexamethasone and High-dose Melphalan in Patients With Relapse After High-dose Melphalan With Autologous Stem Cell Support
Brief Title: Bortezomib and High-dose Melphalan at Myeloma Relapse
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nordic Myeloma Study Group (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Peter Gimsing, Nordic Myeloma Study Group, Rigshospitalet
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMSG 16-07; EudraCT nr 2006-007022-64; KF 02 2006-7206; LMS 2612-3390
Record Dates: First submitted 2007-07-26; First posted 2007-07-27 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Multiple Myeloma
Keywords: high-dose melphalan; bortezomib; response; toxicity; relapse
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bortezomib — 1.3 mg/sqm days -5 and -2 in connection with high-dose melphalan (200mg/sqm day -2) and autologous stem cell support
  Other Names: Velcade

SUMMARY:
The prognosis after retreating with high-dose melphalan with stem cell support after first relapse after high-dose treatment is dependent on the time to first relapse. Bortezomib can increase chemosensitivity of e.g. melphalan. The trial aims at determining the toxicity of adding bortezomib to high-dose melphalan with stem cell support and evaluating whether the time to a second relapse can be prolonged.

DETAILED DESCRIPTION:
Patients with multiple myeloma who have their first treatment demanding relapse after an initial treatment with high-dose melphalan with autologous stem cell support and who have more than 2.0 x 10^6 CD34+ stem cells pr kg bodyweight in the freezer can be included in the trial.

After disease status with basic clinical biochemistry, M-protein in blood and urine, bone marrow investigation including immunophenotyping and total skeletal x-ray the patients are treated with three courses of standard bortezomib (1.3 mg/sqm Days 1,4,8,11) and dexamethasone 20 mg days 1,2,4,5,8,9,11,12. Within 4 weeks the patients receive bortezomib days -5 and -2, high-dose melphalan (200 mg/sqm) day -2, and subsequent at least 2.0 x 10^6 CD34+ stem cells pr kg body weight.

The first month after high-dose therapy the patients are followed closely for toxicity according to the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE), Version 3.0.

The patients are evaluated for response according to EBMT criteria and for event (death or progressive disease).

ELIGIBILITY:
Inclusion Criteria:

* First relapse after ASCT
* Symptomatic myeloma
* More than 2,0 x 10^6 CD34+ stem cells / kg bodyweight in the freezer for stem cell support
* Signed informed consent given prior to any study related activities have been performed
* Age > 18 years

Exclusion Criteria:

* Allogeneic transplantation scheduled as a part of the treatment
* Expected survival of less than one month.
* Performance status (WHO) > 3
* Neuropathy > Grade 3 (neurological symptoms interfering with ADL)
* Non-secreting myeloma
* Other concurrent disease making bortezomib treatment unsuitable
* Positive pregnancy test (only applicable for women with childbearing potential)
* Has known or suspected hypersensitivity or intolerance to melphalan, dexamethasone, boron, mannitol, or heparin, if an indwelling catheter is used
* Uncontrolled or severe cardiovascular disease including myocardial infarction within 6 months of enrolment, New York Heart Association (NYHA) Class III or IV heart failure (Attachment 6, NYHA Classification of Cardiac Disease), uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis
* History of hypotension or has decreased blood pressure (sitting systolic blood pressure [SBP] <= 100 mmHg and/or sitting diastolic blood pressure [DBP] <= 60 mmHg)
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Have received an experimental drug or used an experimental medical device within 4 weeks prior to inclusion into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-06 (Actual); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Comparison of the event free survival after first high-dose melphalan with stem cell support (ASCT) and a second ASCT combined with bortezomib treatment of first relapse | 3 years

SECONDARY OUTCOMES:
Determining the toxicity of bortezomib as part of the high-dose melphalan conditioning | 3 years
Response rate of the second ASCT | 3 years
Marrow regeneration | 3 years
OS compared with the OS of matched controls from the former NMSG | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gimsing, M.D., Principal Investigator — Department of Haematology, Rigshospitalet
Locations (9):
- Denmark (4):
  - Department of Haematology B, Aalborg Hospital, University of Aarhus, Aalborg
  - Dept. of Haematology, Århus University Hospital, Aarhus
  - Department of Haematology, Herlev University Hospital, Herlev
  - Department of Haematology X, Odense University Hospital, Odense
- Norway (3):
  - Hematologisk seksjon, med avd, Haukeland Universitetssykehus, Bergen
  - Department of Hematology, Rikshospitalet, Oslo
  - Hematologisk seksjon, St.Olav Hospital, Trondheim
- Sweden (2):
  - Department of Hematology, Sahlgrenska Sjukhuset, Gothenburg
  - University Hospital Lund, Lund